CLINICAL TRIAL: NCT02657148
Title: A Prospective Observational Clinical Trial to Compare the Effect of Immediate Postpartum Nexplanon Placement Versus Standard Postpartum Contraceptive Care on Consistent Contraceptive Use and Rapid Repeat Pregnancy in Opioid Dependent Women.
Brief Title: Immediate Postpartum Nexplanon Placement in Opioid Dependent Women
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Elizabeth Krans, MD, Assistant Professor, Department of Obstetrics, Gynecology & Reproductive Sciences, University of Pittsburgh
Other Study IDs: PRO15070357; IIS#53505 (Other Grant/Funding Number: Merck Women's Health MISP-RC)
Record Dates: First submitted 2015-09-21; First posted 2016-01-15 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Opiate Addiction; Pregnancy; Contraceptive Behavior; Sexual Behavior
MeSH Terms: conditions — Opioid-Related Disorders; Contraception Behavior; Sexual Behavior | interventions — etonogestrel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Immediate postpartum Nexplanon: Participants who choose to enroll in the immediate postpartum Nexplanon arm will have a etonogestrel contraceptive implant (68 mg) (Nexplanon) placed in the immediate postpartum period (2-4 days following delivery), prior to hospital discharge.
  Interventions: Drug: Nexplanon (etonogestrel contraceptive implant)
- Control: Participants who choose to enroll in the control arm will receive standard postpartum contraceptive care: condoms, Depo Provera (DMPA) or progestin-only pills initiated at any time after delivery, Nexplanon insertion at > 4 weeks after delivery, combined hormonal contraception (e. g. pills, patch, ring) initiated at any time > 4 weeks after delivery or levonorgestrel-intrauterine system or copper IUD insertion any time > 6 weeks after delivery.
  Interventions: Drug: Standard postpartum contraceptive care

INTERVENTIONS:
Drug: Nexplanon (etonogestrel contraceptive implant) — Nexplanon is a single, radiopaque, rod-shaped implant, containing 68 mg etonogestrel indicated for postpartum contraceptive use by women to prevent pregnancy. Nexplanon is designed to be effective for 3 years.
  Other Names: Nexplanon
  Groups: Immediate postpartum Nexplanon
Drug: Standard postpartum contraceptive care — Condoms, Depo Provera (DMPA) or progestin-only pills initiated at any time after delivery, Nexplanon insertion at > 4 weeks after delivery, combined hormonal contraception (e. g. pills, patch, ring) initiated at any time > 4 weeks after delivery or levonorgestrel-intrauterine system or copper IUD insertion any time > 6 weeks after delivery.
  Other Names: Postpartum contraception
  Groups: Control

SUMMARY:
The investigators have designed a single site, Phase IV open label, prospective observational clinical trial to compare the effect of immediate postpartum Nexplanon placement (IPP) versus standard postpartum contraceptive care (control) on consistent contraceptive use and rapid repeat pregnancy at 12 months postpartum in 200 opioid dependent (OD) women.

DETAILED DESCRIPTION:
Background: Opioid dependence in pregnancy has increased dramatically in the last decade. Over 86% of pregnancies conceived by OD women are unintended, compared to 31-43% of pregnancies in the general population. In evaluations of contraceptive use among sexually active women in opioid treatment programs, 40-75% of sexually active OD women report no contraceptive use. Even among women using contraception, 45-55% report using only condoms without more effective, hormonal contraception. Pregnancy and the postpartum period are unique opportunities to provide contraceptive education and services. Long-acting reversible contraception (LARC) has been shown to more effectively prevent rapid repeat, unintended pregnancies compared to other postpartum contraceptive options and does not incur the risk of venous thromboembolism associated with estrogen-containing methods (i.e. pills, ring, patch). No studies have evaluated the impact of immediate postpartum etonogestrel implant (Nexplanon) placement on reproductive health outcomes in OD women, a population at significant risk for rapid repeat, unintended pregnancy. In contrast to an intrauterine device (IUD), Nexplanon is safe to insert regardless of labor and delivery circumstances, does not incur an increased risk of postpartum expulsion and is long-acting, which makes it the ideal contraceptive for the immediate postpartum period.

Study site:This single site study will be conducted at Magee-Womens Hospital (MWH) of the University of Pittsburgh Medical Center.

Study Procedures: Recruitment - participants will be recruited during the third trimester of pregnancy (≥ 28 weeks gestation) during prenatal care visits.

Immediate postpartum Nexplanon placement (IPP) - participants who choose to enroll in the IPP Nexplanon arm will have Nexplanon placed in the immediate postpartum period (2-4 days following delivery), prior to hospital discharge.

Standard postpartum contraceptive care (control) - participants who choose to enroll in the control arm will receive a contraceptive method of their choice according to standard clinical protocols. Standard clinical protocols include condoms, Depo Provera (DMPA) or progestin-only pills initiated at any time after delivery, Nexplanon insertion at > 4 weeks after delivery, combined hormonal contraception (e. g. pills, patch, ring) initiated at any time > 4 weeks after delivery or levonorgestrel-intrauterine system or copper IUD insertion any time > 6 weeks after delivery.

Study Duration: 12 months

ELIGIBILITY:
Inclusion Criteria: Pregnant women, 18 years or older, who meet DSM-V criteria for opioid use disorder confirmed by diagnostic coding in the patient's medical record and/or urinary toxicology screen (UDS) and who plan to deliver at the study site hospital, Magee-Womens Hospital of UPMC (MWH-UPMC).

Exclusion Criteria: Women who have contraindications to etonogestrel use, intrauterine fetal demise or stillbirth, and/or who do not plan to deliver at MWH-UPMC.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women, 18 years or older, who meet DSM-V criteria for opioid use disorder confirmed by diagnostic coding in the patient's medical record and/or urinary toxicology screen (UDS) and who plan to deliver at the study site hospital, Magee-Womens Hospital of UPMC (MWH-UPMC).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Consistent contraception | 12 months postpartum
  Number of participants who use highly effective contraception (all hormonal methods or the copper T380 IUD) for ≥ 80% of the first postpartum year

SECONDARY OUTCOMES:
Rapid, repeat pregnancy | 12 months postpartum
  Number of participants who have a repeat pregnancy within 12 months after delivery
Breastfeeding initiation | 12 months postpartum
  Number of participants who breastfeed after delivery
Postpartum depression | 12 months postpartum
  Edinburgh Postnatal Depression Scale scores
Infant weight gain | 12 months
  Infant weight in kilograms
Infant development | 12 months
  Number of infants that achieve developmental milestones
High-risk sexual behavior | 12 months
  Number of participants who use condoms

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth E Krans, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patrick SW, Schumacher RE, Benneyworth BD, Krans EE, McAllister JM, Davis MM. Neonatal abstinence syndrome and associated health care expenditures: United States, 2000-2009. JAMA. 2012 May 9;307(18):1934-40. doi: 10.1001/jama.2012.3951. Epub 2012 Apr 30. PMID 22546608
- [Background] Heil SH, Jones HE, Arria A, Kaltenbach K, Coyle M, Fischer G, Stine S, Selby P, Martin PR. Unintended pregnancy in opioid-abusing women. J Subst Abuse Treat. 2011 Mar;40(2):199-202. doi: 10.1016/j.jsat.2010.08.011. Epub 2010 Oct 30. PMID 21036512
- [Background] Rabin RF, Jennings JM, Campbell JC, Bair-Merritt MH. Intimate partner violence screening tools: a systematic review. Am J Prev Med. 2009 May;36(5):439-445.e4. doi: 10.1016/j.amepre.2009.01.024. PMID 19362697
- [Background] van Bussel JC, Spitz B, Demyttenaere K. Reliability and validity of the Dutch version of the maternal antenatal attachment scale. Arch Womens Ment Health. 2010 Jun;13(3):267-77. doi: 10.1007/s00737-009-0127-9. Epub 2009 Oct 27. PMID 19859787
- [Background] Brito MB, Ferriani RA, Quintana SM, Yazlle ME, Silva de Sa MF, Vieira CS. Safety of the etonogestrel-releasing implant during the immediate postpartum period: a pilot study. Contraception. 2009 Dec;80(6):519-26. doi: 10.1016/j.contraception.2009.05.124. Epub 2009 Jul 10. PMID 19913145
- [Background] Tocce K, Sheeder J, Python J, Teal SB. Long acting reversible contraception in postpartum adolescents: early initiation of etonogestrel implant is superior to IUDs in the outpatient setting. J Pediatr Adolesc Gynecol. 2012 Feb;25(1):59-63. doi: 10.1016/j.jpag.2011.09.003. Epub 2011 Nov 3. PMID 22051792
- [Background] Grimes DA, Lopez LM, Schulz KF, Van Vliet HA, Stanwood NL. Immediate post-partum insertion of intrauterine devices. Cochrane Database Syst Rev. 2010 May 12;(5):CD003036. doi: 10.1002/14651858.CD003036.pub2. PMID 20464722
- [Background] Tocce KM, Sheeder JL, Teal SB. Rapid repeat pregnancy in adolescents: do immediate postpartum contraceptive implants make a difference? Am J Obstet Gynecol. 2012 Jun;206(6):481.e1-7. doi: 10.1016/j.ajog.2012.04.015. Epub 2012 Apr 16. PMID 22631865
- [Background] Sinha C, Guthrie KA, Lindow SW. A survey of postnatal contraception in opiate-using women. J Fam Plann Reprod Health Care. 2007 Jan;33(1):31-4. doi: 10.1783/147118907779399738. PMID 17389093
- [Background] Gipson JD, Koenig MA, Hindin MJ. The effects of unintended pregnancy on infant, child, and parental health: a review of the literature. Stud Fam Plann. 2008 Mar;39(1):18-38. doi: 10.1111/j.1728-4465.2008.00148.x. PMID 18540521
- [Background] Baldwin MK, Edelman AB. The effect of long-acting reversible contraception on rapid repeat pregnancy in adolescents: a review. J Adolesc Health. 2013 Apr;52(4 Suppl):S47-53. doi: 10.1016/j.jadohealth.2012.10.278. PMID 23535057
- [Background] Morrison CL, Ruben SM, Beeching NJ. Female sexual health problems in a drug dependency unit. Int J STD AIDS. 1995 May-Jun;6(3):201-3. doi: 10.1177/095646249500600311. PMID 7647124
- [Background] Armstrong KA, Kenen R, Samost L. Barriers to family planning services among patients in drug treatment programs. Fam Plann Perspect. 1991 Nov-Dec;23(6):264-6, 270-1. PMID 1786807
- [Background] Ralph N, Spigner C. Contraceptive practices among female heroin addicts. Am J Public Health. 1986 Aug;76(8):1016-7. doi: 10.2105/ajph.76.8.1016. PMID 3728758
- [Background] Armstrong KA, Kennedy MG, Kline A, Tunstall C. Reproductive health needs: comparing women at high, drug-related risk of HIV with a national sample. J Am Med Womens Assoc (1972). 1999 Spring;54(2):65-70, 78. PMID 10319594
- [Background] Black KI, Stephens C, Haber PS, Lintzeris N. Unplanned pregnancy and contraceptive use in women attending drug treatment services. Aust N Z J Obstet Gynaecol. 2012 Apr;52(2):146-50. doi: 10.1111/j.1479-828X.2012.01413.x. Epub 2012 Feb 15. PMID 22335489